CLINICAL TRIAL: NCT04819711
Title: Addressing Perinatal Depression in Deprived Areas of Istanbul, Turkey: a Pilot Randomised Controlled Trial
Brief Title: Addressing Perinatal Depression in Deprived Areas of Istanbul, Turkey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perran Boran (Other)
Collaborators: Medical Research Council (Other Government)
Responsible Party: Sponsor-Investigator, Perran Boran, Professor of Pediatrics, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MR/T038616/1
Record Dates: First submitted 2021-03-25; First posted 2021-03-29 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Perinatal Depression
Keywords: depression; anxiety; disability; sleep; social support
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: two-arm pilot individual randomised controlled trial
Who Masked: Outcomes Assessor
Masking Description: The main outcomes will be recorded by outcome assessors blinded to treatment allocation. It will not be possible to blind antenatal nurses delivering the intervention in participating centres or the participants themselves to intervention allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Thinking Healthy group intervention integrated into antenatal pregnancy school classes
  Interventions: Behavioral: Thinking Healthy Programme
- Control (No Intervention): Participants randomized to the control arm will not be offered the THP intervention but will attend the 5 sessions of the routine group antenatal pregnancy school classes. The class provides education about pregnancy, birth and new-born care and offers support to women. The women will also be able to access all usual care and support offered by the participating hospitals

INTERVENTIONS:
Behavioral: Thinking Healthy Programme — The Thinking Healthy Programme (THP) is an evidence-based intervention that is based on principles of cognitive behavioral therapy. It includes strategies that incorporate behavioral activation, active listening, collaboration with the family, guided discovery, and homework. The adapted THP consists of 5 integrated sessions. Session 1 introduces the programme and focuses on engagement of participants, introduction of THP, and breathing exercises. Session 2 focuses on psychoeducation and problem solving. Session 3 focuses on the mother's well-being and introduces activities such as physical exercises, good sleep practices and ensuring a balanced diet. Session 4 focuses on the mother's relationship with the unborn baby. Session 5 focuses on activating social support from family, friends and peers and provides closure of therapy.
  Arms: Intervention

SUMMARY:
In Turkey, the prevalence rate of perinatal depression has been estimated between 20%-40%, reflecting the global average of 25%. Untreated perinatal depression is of concern not only because of its effect on maternal health but also from the effect that impaired maternal role fulfilment has on the mother-infant bonding and child care and the long-term impact on the infant's physical and cognitive development. Thinking Healthy Programme (THP) is an evidence-based intervention incorporated into the World Health Organization's flagship Mental Health Gap Action Programme, tailored to the perinatal period that has been shown to be effective for depressed or stressed mothers. Turkey prioritize antenatal care, and this provides an opportunity to integrate mental health care into an existing antenatal care programme. Public hospitals operate 'antenatal pregnancy schools' where women are invited to attend 5 weekly group sessions that incorporate education about pregnancy and newborn care. We have developed an on-line group version of the Thinking Healthy Programme which has been designed to be integrated into the routine on-line antenatal pregnancy classes. The intervention has been designed so it is suitable for all women (universal) rather than depressed mothers only (targeted).

The aim of this study is to pilot this adapted on-line group intervention in selected hospitals' pregnancy schools.

The study will be a two-arm pilot individual randomised controlled trial comparing the Thinking Healthy group intervention integrated into antenatal pregnancy school classes with antenatal pregnancy school classes alone. Our sample size of 60 pregnant women (that is 30 participants in each arm of the pilot trial), who are over 18 years old, between 12-30 weeks' gestation, and intend to attend all 5 sessions of the online antenatal classes. Participants in both arms will be assessed for depression and anxiety symptoms, levels of disability, quality of sleep, perceived social support, coping skills, and relationship with partner. All one hundred and twenty women will get a detailed assessment initially and 4-6 weeks after the intervention. Some of the study participants and antenatal nurses delivering these sessions will be approached for in-depth qualitative interviews to explore the acceptability, feasibility and perceptions of the study participants' receiving the intervention sessions.

DETAILED DESCRIPTION:
Systematic reviews provide robust evidence that perinatal depression can be treated effectively in low to middle income countries with psychological treatments delivered by non-specialists. The intervention with the strongest demonstrated effect size is the Thinking Healthy Programme, the first psychological intervention to be incorporated into the World Health Organization's flagship Mental Health Gap Action Programme (mhGAP). Turkey prioritize antenatal care, and this provides an opportunity to integrate mental health care into an existing antenatal care programme.

Public hospitals operate 'antenatal pregnancy schools' where women are invited to attend 5 weekly group sessions that incorporate education about pregnancy and newborn care. The groups usually consist of 8-10 mothers and are run by antenatal nurses. During the COVID19 pandemic, these classes have been adapted into an on-line platform. Group interventions are less resource-intensive per person helped than individual interventions and are possibly more cost-effective. We have developed an on-line group version of the Thinking Healthy Programme which has been designed to be integrated into the routine on-line antenatal pregnancy classes. The intervention has been designed so it is suitable for all women (universal) rather than depressed mothers only (targeted).

Our objectives are to conduct a pilot/feasibility study of the on-line group intervention in a socioeconomically deprived population in Istanbul, Turkey.

The primary aim of this pilot study is not to test a specific hypothesis but to:

1. test all operational elements including: the acceptability and feasibility of the intervention including training and supervision; the materials developed such as the manual, visual aids, and added activities to promote perinatal mental health and psychosocial well-being;
2. test the willingness of women, and antenatal nurses to participate (recruitment rates), respond to questionnaires, and be followed up (attrition rates); and
3. test the procedures for outcome measures as well as training and supervision. Quantitative methods will closely follow the procedures for a future definitive trial. The results will be used to finalise the intervention content and structure, to establish appropriate support systems, and to finalize all materials.

The study will be conducted in socioeconomically deprived districts of Istanbul within the catchment area of the First Region of the Public Hospitals Union. Primary institution will be Marmara University Hospital which has an affiliation with the Ministry of Health. With the support of Turkish Ministry of Health, the hospital operates 'antenatal pregnancy schools'.

Our study participants will include all consecutive pregnant women who have been offered, and accepted to attend, the on-line antenatal care classes during the study recruitment period.

Because this is a feasibility/pilot trial, sample size calculations have not been conducted. Our sample size of 60 (that is 30 participants in each arm of the pilot trial) is based on the pragmatics of recruitment and the necessities for examining feasibility. The intervention and control arms will each consist of 3 groups per arm with 10 participants per group, respectively.

The research design is a two-arm pilot individual randomised controlled trial comparing the Thinking Healthy group intervention integrated into antenatal health classes with antenatal health classes alone.The unit of randomization for the pilot trial will be individuals (i.e, eligible pregnant women). The generation of random allocation sequence will be carried-out by an independent person at the University of Liverpool UK (not involved in the enrolment of participants into the trial). Simple random numbers will be generated and the case will be assigned a Trial Number and treatment allocation (TAU or THP) which will be emailed back to the Local PI at Marmara in an encrypted form who will be responsible for notifying the site coordinator. The site coordinator will then inform both the participants and the designated nurses for the particular treatments to commence. To minimise the threat of selection bias through allocation concealment, the team recruiting/enrolling participants will be separate to the team opening the encrypted forms and informing participants about the treatment that will receive.

The main outcomes will be recorded by outcome assessors blinded to treatment allocation. Participants will be asked before the interview with the assessor not to reveal anything about their sessions. The outcome assessors will not have information about the on-line groups. It will not be possible to blind therapists and antenatal nurses in participating centres or the participants themselves to intervention allocation.

Intervention The Thinking Healthy Programme (THP) is an evidence-based intervention that is based on principles of cognitive behavioral therapy. It includes strategies that incorporate behavioral activation, active listening, collaboration with the family, guided discovery, and homework. THP was designed to be delivered by community health workers, and it was the first low-intensity psychological intervention to be adopted by WHO. THP has been translated and adapted into Turkish. For the current study, we have developed an on-line group version of the Thinking Healthy Programme which has been designed to be integrated into the routine on-line antenatal pregnancy classes. It will be delivered by trained antenatal nurses who routinely run the antenatal classes. The routine on-line antenatal classes consist of 5 weekly group sessions that incorporate education about pregnancy and new-born care. The groups usually consist of 8-10 mothers. Our adapted 'group' version of the Thinking Healthy Programme will be incorporated into these antenatal pregnancy classes. The adapted THP consists of 5 integrated sessions. Session 1 introduces the programme and focuses on engagement of participants, introduction of THP, and breathing exercises. Session 2 focuses on psychoeducation and problem solving. Session 3 focuses on the mother's well-being and introduces activities such as physical exercises, good sleep practices and ensuring a balanced diet. Session 4 focuses on the mother's relationship with the unborn baby. Session 5 focuses on activating social support from family, friends and peers and provides closure of therapy.

Participants randomized to the control arm will not be offered the THP intervention but will attend the 5 sessions of the routine group antenatal class. The class provides education about pregnancy, birth and new-born care and offers support to women. The women will also be able to access all usual care and support offered by the participating hospitals.

Assessments will take place at baseline on recruitment and one month after conclusion of the intervention sessions.

Procedures for human subjects' protection in this research will follow guidelines and policies of the Institutional Reviews Boards (IRBs) of the sponsoring organization, the University of Liverpool and the implementing partner, University of Marmara, School of Medicine.

The data and safety monitoring plan will involve the continuous evaluation of safety, data quality and data timeliness. Incoming data will be cleaned and compiled on a regular basis and examined for unusual or unexpected patterns. PIs and project coordinators will conduct continuous review of data and participant safety at monthly Project Management Group meetings and the discussion will be documented in minutes. The governance mechanisms will provide oversight to the programme. The governance and administrative activities will be based in Istanbul at Marmara University (School of Medicine) and will be the responsibility of the site investigators.

Flow of participants through the trial will be presented as the trial flow chart. Descriptive statistics including socio-demographic characteristics and all baseline measures across arms will be tabulated to check for any baseline imbalances among the participants. Mean and standard deviation scores for all continuous measures shall be presented, followed by univariate associations between demographic variables and severity of symptoms. While the study is not powered to test any hypothesis, exploratory intention to treat analysis will be conducted to compare the two treatment groups. For baseline comparisons, t-tests will be conducted for continuous variables and chi-squared test for categorical ones. At follow up, comparisons will be made using analysis of covariance with baseline score as a co-variate. Any significant baseline imbalances will be treated as co-variates and adjusted for in analysis. All qualitative data will be analysed using framework analysis approach

ELIGIBILITY:
Inclusion Criteria:

* pregnant women over 18 years between 12-30 weeks' gestation have access to internet, intend to attend all 5 sessions of the antenatal classes

Exclusion Criteria:

* currently receiving any form of counselling or mental health care, who report suicidal ideation women who have a miscarriage, stillbirth or preterm birth will also be excluded from the follow-up assessment

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women between 12-30 weeks' gestation
Enrollment: 88 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2021-10-20 (Actual); Study Completion 2021-11-11 (Actual)

PRIMARY OUTCOMES:
Change in Depression | Baseline and at 4-6 weeks after the intervention
  Edinburgh Postnatal Depression Scale. This is a 10-item self-administered scale, each item is rated on a four-point scale, giving maximum scores of 30. A score of 13 or more is considered to be a significant case of postnatal depression, while scores of 10 to 12 represent borderline. It is developed for detection of symptoms of psychosocial distress during pregnancy and in the postnatal period.

SECONDARY OUTCOMES:
Change in Disability | Baseline and at 4-6 weeks after the intervention
  WHO Disability Assessment Schedule. WHODAS 2.0 covers six domains (cognition, mobility, self-care, getting along, life activities and participation), and assesses difficulties people have during the last 30 days. Difficulties are scored on a five-point Likert scale as none, mild, moderate severe or extreme. WHODAS 2.0 has been validated cross-culturally
Change in Depression | Baseline and at 4-6 weeks after the intervention
  Patient Health Questionnaire-9. Patient Health Questionnaire (PHQ-9) is a nine item instrument which can diagnose as well as measure severity[17]. As a severity measure, the PHQ-9 score ranges from 0 to 27, with each of the nine items scored from 0 (not at all) to 3 (nearly every day). A score of 10 or above indicates Depressive disorder.
Change in Anxiety | Baseline and 4-6 weeks after the intervention
  Generalised Anxiety Disorder questionnaire (GAD-7). The questionnaire score is calculated by assigning scores of 0, 1, 2, and 3, to the response categories of 'not at all', 'several days', 'more than half the days', and 'nearly every day', respectively, and adding together the scores for the seven questions. Scores of 5, 10, and 15 are taken as the cut-off points for mild, moderate and severe anxiety, respectively.
Change in Sleep quality | Baseline and 4-6 weeks after the intervention
  Pittsburgh Sleep Quality Index (PSQI). It was developed to evaluate sleep quality in clinical studies. The items in the PSQI were arranged using clinical observations of patients with sleep disorders, other scales about sleep quality specified in the literature, and an 18-month clinical observation period regarding PSQI. If the PUKI global score is greater than 5, it indicates poor sleep quality
Change in Perceived social support | Baseline and 4-6 weeks after the intervention
  Multidimensional Scale of Perceived Social Support (MSPSS). The scale will be used to understand the changes in perceived social support. The MSPSS is a 12-item scale designed to measure perceived social support from three sources: Family, Friends, and a Significant Other. It has 12-item and every item uses a seven-point Likert scale ranging from 1 (very strongly disagree) to 7 (very strongly agree). A higher score indicates greater the social support perceived by an individual; the total possible score ranges 12~84, or it can be scored according to its subscales by adding the items in each subscale and then dividing by 4.
Change in Coping skills | Baseline and 4-6 weeks after the intervention
  Brief-COPE. Change in coping skills will be assessed by the Brief-COPE which is a 28 item self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. The Brief-Cope was developed as a short version of the original 60-item COPE scale, which was theoretically derived based on various models of coping. "Coping" is defined broadly as an effort used to minimize distress associated with negative life experiences. The scale can determine someone's primary coping styles as either Approach Coping, or Avoidant Coping. In addition, the following subscales are reported: Self-distraction, Active coping, Denial, Substance use, Use of emotional support, Use of instrumental support, Behavioral disengagement, Venting, Positive reframing, Planning, Humor, Acceptance, Religion, & Self-blame.
Change in relationship with partner | Baseline and 4-6 weeks after the intervention
  Relationship Assessment Scale (RAS). This is a 7 item scale, used to assess subjective satisfaction with a given relationship. Answers are rated on a 5 point Likert scale, ranging from 1 (not well), to 5 (very well). The respondent's average score is obtained after reverse scoring items 4 and 7. Although this scale was originally created to assess romantic relationships, created a generic version that they found to be sufficiently reliable: Cronbach's α = .89 for parents, .87 for friends, and .90 for romantic partners.

CONTACTS AND LOCATIONS:
Locations (2):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)
- University of Liverpool, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Requests for wider sharing of data (for example in response to information on the UoL, Marmara University webpages and in publications about the study and willingness to share), will be addressed on a case-by-case basis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: when data is ready for analysis
Access Criteria: Any data sharing request will be made to investigators through a pre-defined data requisition form. This form will contain information about the applicant, institution, purpose of data request, study objectives, ethical clearance of the study, etc. Once a request has been made the data governance body will discuss if that request was appropriate and meets the criteria set by the participating centres; data will be released following signing of the data sharing agreement. The data will be stored on the Marmara University and UoL servers and not be deposited in any 'community' database.

REFERENCES:
- [Derived] Boran P, Donmez M, Baris E, Us MC, Altas ZM, Nisar A, Atif N, Sikander S, Hidiroglu S, Save D, Rahman A. Delivering the Thinking Healthy Programme as a universal group intervention integrated into routine antenatal care: a randomized-controlled pilot study. BMC Psychiatry. 2023 Jan 6;23(1):14. doi: 10.1186/s12888-022-04499-6. PMID 36604685